CLINICAL TRIAL: NCT06649019
Title: Evaluation of Lens Rotation in Habitual Wearers of Toric, Soft Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-6576
Record Dates: First submitted 2024-10-16; First posted 2024-10-18 (Actual); Results first posted 2026-01-07 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- AO1DfA/DT1fA (Experimental): Eligible subjects will be randomized into the AO1DfA/DT1fA wear sequence, to wear the test lens followed by the control lens, bilaterally, with a 1-to-10 day(s) washout period between wear periods.
  Interventions: Device: ACUVUE OASYS 1-Day for Astigmatism (AO1DfA); Device: Dailies Total 1 for Astigmatism (DT1fA)
- DT1Fa/AO1DfA (Experimental): Eligible subjects will be randomized into the DT1Fa/AO1DfA wear sequence, to wear the control lens followed by the test lens, bilaterally, with a 1-to-10 day(s) washout period between wear periods.
  Interventions: Device: ACUVUE OASYS 1-Day for Astigmatism (AO1DfA); Device: Dailies Total 1 for Astigmatism (DT1fA)

INTERVENTIONS:
Device: ACUVUE OASYS 1-Day for Astigmatism (AO1DfA) — Test Lens
Device: Dailies Total 1 for Astigmatism (DT1fA) — Control Lens

SUMMARY:
This will be a single site, 2-visit, randomized, controlled, single-masked, non-dispensing, bilateral wear, 2x2 cross over study to assess visual acuity.

ELIGIBILITY:
Inclusion Criteria:

Potential subjects must satisfy all of the following criteria to be enrolled in the study:

1. Read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
3. Be between 18 and 39 years of age (inclusive) at the time of screening.
4. Habitually wear soft, toric contact lenses in both eyes in a daily or daily disposable wear modality (i.e. not extended wear modality). Habitual wearer is defined as a minimum of 6 hours per day, for a minimum of 2 days per week during the past 30 days.
5. Possess a wearable pair of spectacles that provide correction for distance vision (if applicable).
6. Have the spherical component of their vertex-corrected distance refraction within the range +4.00 to -6.00 DS (inclusive) in both eyes.
7. Have the magnitude of the cylindrical component of their vertex-corrected distance refraction between 0.75 DC and 2.50 DC in both eyes.
8. Have best corrected monocular distance visual acuity of 0.2 or better in each eye.

Exclusion Criteria:

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

1. Be currently pregnant or lactating.
2. Be diabetic.
3. Be currently using any ocular medications or have any ocular infection of any type.
4. By self-report, have any ocular or systemic disease, allergies, infection, or use of medication that might contraindicate or interfere with contact lens wear, or otherwise compromise study endpoints, including infectious disease (e.g., hepatitis, tuberculosis), contagious immunosuppressive disease (e.g., Human Immunodeficiency Virus [HIV]), autoimmune disease (e.g. rheumatoid arthritis, Sjögren's syndrome), or history of serious mental illness or seizures. See section 9.1 for additional details regarding excluded systemic medications.
5. Have habitually worn rigid gas permeable (RGP) lenses, orthokeratology lenses, or hybrid lenses (e.g. SynergEyes, SoftPerm) within the past 6 months.
6. Be currently wearing monovision or multifocal contact lenses.
7. Be currently wearing lenses in an extended wear modality.
8. Be currently wearing or have had worn Acuvue® Oasys 1-Day for Astigmatism, or Dailies® Total1 for Astigmatism lenses during the last 3 months.
9. Have a history of strabismus or amblyopia.
10. Be an employee (e.g., Investigator, Coordinator, Technician) or immediate family member of an employee (including partner, child, parent, grandparent, grandchild or sibling of the employee or their spouse) of the clinical site.
11. Have participated in a contact lens or lens care product clinical trial within 7 days prior to study enrollment.
12. Have clinically significant (grade 3 or higher on the Efron grading scale) slit lamp findings (e.g., corneal edema, neovascularization or staining, tarsal abnormalities or bulbar injection) or other corneal or ocular disease or abnormalities that contraindicate contact lens wear or may otherwise compromise study endpoints (including entropion, ectropion, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, moderate or above corneal distortion, herpetic keratitis).
13. Have fluctuations in vision due to clinically significant dry eye or other ocular conditions.
14. Have had or have planned (within the study period) any ocular or intraocular surgery (e.g., radial keratotomy, PRK, LASIK, iridotomy, retinal laser photocoagulation, etc.).

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2024-12-06 (Actual); Primary Completion 2024-12-16 (Actual); Study Completion 2024-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Vision Care, Inc. Clinical Trial, Study Director — Johnson & Johnson Vision Care, Inc.
Locations (1):
- The University of Manchester, Department of Optometry & Neuroscience, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 6 subjects were enrolled at a single clinical site. Of those enrolled, 1 subject failed to meet all eligibility criteria and 5 subjects were dispensed both study lenses and completed the study.
Groups:
- Delefilcon A/Senofilcon A: Subjects that wore the delefilcon A lens in the first period and senofilcon A in the second period.
- Senofilcon A/Delefilcon A: Subjects that wore the senofilcon A lens in the first period and the delefilcon A lens in the second period.
Period: Period 1
Arm/Group | Delefilcon A/Senofilcon A | Senofilcon A/Delefilcon A
Started | 2 | 3
Completed | 2 | 3
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Delefilcon A/Senofilcon A | Senofilcon A/Delefilcon A
Started | 2 | 3
Completed | 2 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects dispensed a study lens.
Groups:
- All Dispensed Subjects: All subjects dispensed a study lens
Arm/Group | All Dispensed Subjects
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.6 (5.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 5

OUTCOME MEASURES:

1. Primary Outcome: Distance Monocular Visual Acuity (LogMAR)
Description: Distance visual acuity was measured monocularly at 6 meters after lens fitting under high-luminance high contrast (HLHC) lighting conditions using the Eurolens computerized logMAR VA chart. Lower scores indicate better visual acuity. A value of 0.0 logMAR is equivalent to 20/20 vision on a Snellen visual acuity chart.
Time Frame: Approximately 15-minutes Post Lens Insertion
Population: All subjects fitted both study lenses and completed the study
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: Eyes
Groups:
- Senofilcon A: Subjects that wore the senofilcon A lens in either the first or second period.
- Delefilcon A: Subjects that wore the delefilcon A lens in either the first or second period.
Arm/Group | Senofilcon A | Delefilcon A
Number analyzed (Participants) | 5 | 5
Number analyzed (Eyes) | 10 | 10
logMAR | -0.07 (0.084) | -0.07 (0.050)

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study; approximately 1-10 days per subject.
Description: All subjects fitted at least 1 study lens.
Arm/Group | Senofilcon A | Delefilcon A
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-10-03): https://cdn.clinicaltrials.gov/large-docs/19/NCT06649019/Prot_SAP_001.pdf